CLINICAL TRIAL: NCT04160507
Title: Duke APOL1 Research Biorepository
Acronym: DARB
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00103657
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: End Stage Kidney Disease
Keywords: ESKD; APOL 1 gene; Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases | interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMCs) will be isolated from the blood using standard Ficoll-Paque technique. A fraction of the PBMCs will be cryopreserved and stored at for future analysis. We will submit a separate IRB protocol for use of future unspecified research with these samples. The remaining fraction of PBMCs will be used to generate inducible pluripotentent stem cells (iPSCs). These iPSC would be differentiated into kidney cells which could then be further studied. While no plans exist to immortalize any of these cell lines, the consent form does allow for creating immortalized cell lines in the future. Residual plasma will also be stored separately for additional analysis. Kidney cells shed into urine would also be a potential source of iPSCs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy black adults 50 and over: Healthy black adults age 50 and over with no known history of kidney disease will be recruited as controls in this study.
  Interventions: Other: Biorepository
- black adult cases with non-diabetic nephropathy: black adult cases with non-diabetic nephropathy
  Interventions: Other: Biorepository

INTERVENTIONS:
Other: Biorepository — To collect and store biological samples (whole blood and urine), along with relevant medical information, from adult inpatients and outpatients. Buffy coats will also be received from H3Africa Kidney Disease Research Network.

SUMMARY:
The Duke ApoL1 Nephropathy Biorepository aims to address needs within non-diabetic kidney failure research by utilizing existing and, when necessary, developing new infrastructure to support the consent of patients and the collection of dedicated samples for ApoL1 Nephropathy biorepository.

The mutations in ApoL1 gene that are strongly associated with kidney disease are only present in individuals of recent African ancestry (i.e., black people). Caucasians do not have these ApoL1 mutations nor the associated kidney disease. Therefore, majority of subjects recruited for this study will be self-identified African Americans, Afro-Caribbean and other black individual. Study subjects will include individuals with end stage kidney disease and those without any clinical evidence of kidney disease.

Additionally, healthy black adults with no known history of kidney disease will be recruited as controls in this study because they are the only group that can fill this role.

DETAILED DESCRIPTION:
The risk of end stage kidney failure among African Americans is 4 times that of Caucasian Americans. This excess risk of kidney failure is largely attributable to mutations in apolipoprotein L1 gene. While 10-15% of African Americans in the United States possess kidney disease-associated ApoL1 mutations, nearly 40% of African Americans on dialysis have these mutations. There are significant gaps in the understanding of the pathophysiology of ApoL1-nephropathy. Only some of the people with ApoL1 mutations develop kidney failure. The pathways that link ApoL1 mutations with end stage kidney failure are not understood. Because kidney biopsy is generally obtained from patients with evidence of kidney disease-whose kidneys have experienced significant damage and sclerosis-access to the relevant kidney cells is very limited. However, recent advancements in biomedical research have made it possible to develop kidney-like cells from inducible pluripotent stem cells (iPSCs) which were derived from blood cells of individuals. This innovative technique will allow us to generate iPSC-derived cells from the blood of individuals who have developed ApoL1-nephropathy for the purpose studying them in research lab so as to decipher the cellular mechanism of their kidney failure.

ELIGIBILITY:
Inclusion Criteria:

* Majority of subjects recruited for this study will be self-identified African Americans, Afro-Caribbean and other black individuals. Study subjects will include individuals at various stages of kidney disease and those without any clinical evidence of kidney disease.
* Healthy black adults, age 50 and older with no known history of kidney disease will be recruited as controls

Exclusion Criteria:

* Black adult cases with diabetic nephropathy
* Healthy controls with kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mutation in ApoL1 gene is associated with increased risk of non-diabetic kidney disease in individuals of recent African descent-i.e., only black people are affected. Therefore, black adult cases with non-diabetic nephropathy or healthy controls aged 18 years or older will be recruited for consent into the DANB.
  Caucasians do not have these ApoL1 mutations nor the associated kidney disease. Therefore, majority of subjects recruited for this study will be self-identified African Americans, Afro-Caribbean and other black individual. Study subjects will include individuals at various stages of kidney disease and those without any clinical evidence of kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Biorepository | 5 years
  Number of biological samples collected and stored (whole blood and urine).

SECONDARY OUTCOMES:
Future study samples | 5 years
  1) Number of biological samples for future studies, including epigenetic and biomarker research.

OTHER OUTCOMES:
Understanding the mechanisms by which mutations in ApoL1 gene cause kidney disease, including identification of cellular and epigenetic risk factors | 5 years
  Number of biological samples to understand the mutations in ApoL1

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share IPD data with other researchers.